CLINICAL TRIAL: NCT03433976
Title: Comparison of the Duration of Motor Block After Spinal Anesthesia for Planned Cesarean Sections: Hyperbaric Prilocaïne Versus Hyperbaric Bupivacaine
Brief Title: Prilocaine or Bupivacaine for Spinal Anesthesiain Pregnant
Acronym: Césarcaïne
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hopital Saint Roch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UF9859
Record Dates: First submitted 2017-12-21; First posted 2018-02-15 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-03

CONDITIONS: Cesarean
Keywords: Caesarean section; spinal anesthesia; Prilocaïne; motor block
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Bupivacaine (Other): spinal anesthesia for planned cesarean sections control group
  Interventions: Drug: spinal anesthesia
- Hyperbaric Prilocaïne (Active Comparator): spinal anesthesia for planned cesarean sections
  Interventions: Drug: spinal anesthesia

INTERVENTIONS:
Drug: spinal anesthesia — spinal anesthesia for planned cesarean sections

SUMMARY:
The planned cesarean section is an intervention with a standard operating time of less than 40 minutes in trained teams. Hyperbaric Bupivacaine is the local anesthetic (LA) reference for these operations. But the duration of its motor block is generally greater than 3 hours. The purpose of this study is to show a reduction in motor block time with hyperbaric Prilocaine by at least 30 minutes, which would allow mothers and their children to return to the maternity ward earlier and thus improve the circulation of patients within the maternity's PACU.

DETAILED DESCRIPTION:
Prospective study, randomized into two parallel groups (Hyperbaric Prilocaïne versus hyperbaric Bupivacaine), double-blind, monocentric (Clinique Saint Roch in Montpellier).

The number of subjects required is 50 patients, 25 per group.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy
* Scheduled caesarean section
* Non-multiple pregnancy
* Age of patient: 18 years and over
* Height of patient: between 155 and 175 cm
* Affiliated patients or beneficiaries of a Social Security System
* Signature of the patient's consent

Exclusion criteria:

* Patient <18 years
* Pathological pregnancy
* Multiple pregnancy
* Emergency caesarean
* Patients who cannot give informed consent (not French speaking)
* Refusal of the patient
* Contraindications to spinal anesthesia
* Contraindications to Prilocaine
* Contraindications to Bupivacaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-05-07 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
duration of motor block | up to 6 hours
  To compare the duration of motor block after spinal anesthesia with hyperbaric Prilocaïne versus hyperbaric Bupivacaine This evaluation is done every 15 min from the entrance to the recovery room (PACU); the motor block stops being evaluated when the modified bromination score reaches 4

SECONDARY OUTCOMES:
The upper sensory level | 15 minutes after the LA injection
  The upper sensory level obtained 15 minutes after the LA injection
Hypotensive episodes | 1 day
  Hypotensive episodes
The time between injection and incision | 1 day
  The time between injection and incision
The duration of the intervention | 1 day
  The duration of the intervention
The time to return to the standard maternity ward | 1 day
  The time to return to the standard maternity ward
APGAR score of newborns at birth | 1 day
  APGAR score of newborns at birth. L'APGAR Apgar score is a method to quickly summarize the health of newborn children.
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).
  The test is generally done at one and five minutes after birth, and may be repeated later if the score is and remains low. Scores 7 and above are generally normal, 4 to 6 fairly low, and 3 and below are generally regarded as critically low.
The delay between spinal anesthesia and the first emergency analgesic injection | 1 day
  The delay between spinal anesthesia and the first emergency analgesic injection
Assessment of pain (VAS) | 1 day
  Pain on arrival and departure of PACU and at 24 hours. Pain will be assessedby VAS (Visual Analogue Scale); Patients rate pain on VAS from 0-10, 0 being no pain and 10 being the worst pain imaginable..
The delay between spinal anesthesia and the first injection of second-line analgesia | 1 day
  The delay between spinal anesthesia and the first injection of second-line analgesia : delay between spinal anesthesia ans the need of rescue analgesia
The presence of neuro-sensory disorders within 24 hours postoperatively | 1 day
  The presence of neuro-sensory disorders within 24 hours postoperatively
The presence of post lumbar puncture syndrome | 1 day
  The presence of post lumbar puncture syndrome
score de satisfaction | 1 day
  Patient satisfaction score at 24 hours will be assessed by VAS (Visual Analogue Scale); Patients rate satisfaction on VAS from 0-10, 0 being no satisfaction and 10 being total satisfaction
Statifaction of the Surgeon | 1 day
  The surgeon assessed his satisfaction while the cesarien section. The surgeon satisfaction score at 24 hours will be assessed by VAS (Visual Analogue Scale); Surgeon rate satisfaction on VAS from 0-10, 0 being no satisfaction and 10 being total satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: christophe DADURE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Chapron K, Sleth JC, Capdevila X, Bringuier S, Dadure C. Hyperbaric prilocaine vs. hyperbaric bupivacaine for spinal anaesthesia in women undergoing elective caesarean section: a comparative randomised double-blind study. Anaesthesia. 2021 Jun;76(6):777-784. doi: 10.1111/anae.15342. Epub 2021 Jan 11. PMID 33428221